CLINICAL TRIAL: NCT06715085
Title: Multicenter, Randomized, Single-blind, Controlled Clinical Trial to Evaluate the Safety and Efficacy of PRGF-ENDORET® Infiltrations in the Treatment of Low Back Pain.
Brief Title: PRGF-ENDORET® Infiltrations in the Treatment of Low Back Pain.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Biotechnology Institute IMASD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BTIIMD-03-EC-23-DISC
Record Dates: First submitted 2024-11-21; First posted 2024-12-04 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Diseases [C] - Musculoskeletal Diseases [C05
MeSH Terms: interventions — Intercellular Signaling Peptides and Proteins; Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Plasma Rich in Growth Factors (PRGF) (Experimental): The PRGF application consists of three series of infiltrations in the intervertebral disc, epidural space and facets, with a frequency of two weeks.
  Interventions: Drug: Plasma Rich in Growth Factors (PRGF)
- Control: Corticosteroid solution (Celestone Cronodose suspension for injection) in saline solution. (Active Comparator): The corticosteroid solution application consists of two series of infiltrations of solution of corticosteroid (Celestone Cronodose injectable suspension [betamethasone]) and saline solution in the epidural space and in the facets, with a periodicity of one month between them.
  Interventions: Drug: Corticosteroid solution (Celestone Cronodose suspension for injection) in saline solution.

INTERVENTIONS:
Drug: Plasma Rich in Growth Factors (PRGF) — The PRGF application consists of three series of infiltrations in the intervertebral disc, epidural space and facets, with a frequency of two weeks.
  Other Names: PRGF injection
  Arms: Experimental: Plasma Rich in Growth Factors (PRGF)
Drug: Corticosteroid solution (Celestone Cronodose suspension for injection) in saline solution. — The corticosteroid solution application consists of two series of infiltrations of solution of corticosteroid (Celestone Cronodose injectable suspension [betamethasone]) and saline solution in the epidural space and in the facets, with a periodicity of one month between them.
  Other Names: Corticosteroid solution
  Arms: Control: Corticosteroid solution (Celestone Cronodose suspension for injection) in saline solution.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of PRGF in reducing pain and improving patients' quality of life. Researchers will compare an experimental drug (Plasma Rich in Growth Factors) to a control corticosteroid solution in saline solution.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age (≥18 years).
* Patients diagnosed by Magnetic Resonance Imaging (MRI) with lumbar intervertebral disc degeneration(s) (Pfirrmann Scale > 1).Patients with positive signs in MRI at L4-L5 and/or L5-S1 levels, including rupture of the annulus fibrosus, annular fissure, with or without disc herniation in its protrusion form will be included.
* Patients with low back pain with symptoms of low back pain for at least 3 months of evolution that has not responded to drug treatment.
* Numerical pain scale (COMI PAIN SCORE): between 6 and 10, average of the last month.
* Availability of an MRI performed in the last six months to allow the diagnosis.
* Availability of a complete blood test (hemogram, basic biochemistry and coagulation tests) performed in the last two months.
* Signed informed consent to participate in the clinical trial and authorization for data processing by the different centers involved for subsequent scientific publication.

Exclusion Criteria:

* Patients with lumbar fracture, extruded herniated discs and herniated discs with signs of calcification are excluded.
* Patients with severe discopathies at levels adjacent to L4-L5 and/or L5-S1.
* Patients who have previously undergone spinal surgery.
* Patients who have undergone invasive procedures on the spine in the last 6 months, such as infiltrations, blocks, lavage or lumbar rhizolysis.
* Patients with neurogenic motor claudication.
* Patients with severe cardiovascular diseases, central nervous system diseases, epilepsy, coagulopathies, immunological diseases, infectious diseases (e.g. Hepatitis B and C, HIV, Syphilis), cancer or neurodegenerative pathologies.
* Patients with a history of drug use (e.g. alcoholism or others) and mental illness or marked psychological conditions related to pain.
* Morbidly obese patients (BMI > 40 kg/m2).
* Women who are pregnant or breastfeeding or women of childbearing age who are not taking effective contraceptive measures as outlined in the Clinical Trials Facilitation and Coordination Group (CTFG) "Recommendations Regarding Contraception and Pregnancy Testing in Clinical Trials" V 1.1.
* Patients with pathologies that produce marked alterations in the efficacy of PRGF or coagulation, such as, for example: poorly controlled diabetes mellitus (glycosylated hemoglobin above 9%), hematological alterations (thrombopathy, thrombopenia, anemia with Hb < 9), being subjected to immunosuppressive and/or dicoumarinic treatments, or any treatment with systemic corticosteroids during the 6 months prior to inclusion in the study
* Patients who present allergy to any component of the sedation or to the corticoid.
* Patients who have received previous back treatment with PRGF in the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of PRGF in reducing pain and improving patients' quality of life. | 6 moths follow up
  Efficacy: evaluation of the Oswestry Disability Index (ODI) (also known as the Oswestry Low Back Pain Disability Questionnaire).
  1. Pain intensity / 2. Personal care (washing, dressing etc)/ 3. Lifting / 4. Walking /5. Sitting /6. Standing / 7.Sleeping /8. Sex life (if applicable)/9. Social life /10. Travelling
  For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. If all 10 sections are completed the score is calculated as follows:
  Example: 16 (total scored) --> 50 (total possible score) x 100 = 32% Minimum detectable change (90% confidence): 10% points (change of less than this may be attributable to error in the measurement)
  0% to 20%: minimal disability 21%-40%: moderate disability 41%-60%: severe disability 61%-80%: crippled 81%-100%: either bed-bound or exaggerating their symptoms

SECONDARY OUTCOMES:
Percentage of treatment failures at 1, 3, and 12 months follow-up (following the definition in 8.7) | 1, 3, and 12 months follow-up
  Percentage of treatment failures at 1, 3, and 12 months follow-up

OTHER OUTCOMES:
Evaluation of incidence and type of adverse events | Up to 56 weeks
  Safety variables: each of the adverse events will be described, with a frequency analysis of the safety variables by treatment group, and a subsequent comparison of these by means of the chi-square test.
Cost-effectiveness variables | Up to 56 weeks
  Incremental Cost-Effectiveness Ratio (ICER). The two arms of the trial will be compared to estimate the ICER. Costs will be calculated at the individual level and prospectively.
Effectiveness variable | Up to 56 weeks
  As a measure of effectiveness, quality of life adjusted life years (QoLs) will be calculated as a function of the duration measured by the study and the EuroQol values obtained before and at 56 weeks.
Evaluation of the COMI scale. | 1 , 3, and 12 months of follow-up
  Evaluation of the Core Outcome Measures Index (COMI) scale. It is scored from 0 to 10, the lower the score, the better the result.
Evaluation of the SF-12 scale | 1, 3, 6 and 12 moths follow up
  SF-12 Health Survey. This survey asks for the views about health. The result obtained depends on an algorithm. From the physical domain of the scale, the best result is 56.57 and the worst, 23.99. From the mental domain of the scale, the best result is 60.75 and the worst 19.06.
Evaluation of the EQ-5D-5L Survey | 1, 3, 6 and 12 moths follow up
  To assess the quality of life (EQ-5D-5L survey) related to health or perceived health (in its two aspects, physical and mental). Score from 0 to 100 with 100 being the best result in terms of health.
Radiological imaging (MRI) results | 1 year
  Differences at 12 months with respect to baseline determinations of the Pfirrmann grade
Radiological imaging (MRI) results | 1 year
  Differences at 12 months with respect to baseline determinations of the size of the disc herniation.
Radiological imaging (MRI) results | 1 year
  Differences at 12 months with respect to baseline determinations of the Intervertebral space height (endplate to endplace).
Radiological imaging (MRI) results | 1 year
  Differences at 12 months with respect to baseline determinations of the disc volume.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Eduardo Anitua, Vitoria-Gasteiz, Alava, Spain